CLINICAL TRIAL: NCT03520972
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Dose Cohort Study to Evaluate the Efficacy and Safety of Twelve Once-weekly Subcutaneous Doses of PB-119 in Drug-naïve Subjects With Type 2 Diabetes Mellitus
Brief Title: Dose-finding of PB-119 Administered Subcutaneously Once-weekly Versus Placebo in Drug-naïve T2DM Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PB119201
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PB-119 75ug (Experimental): PB-119 injection 75ug subcutaneously injected once-weekly for 12 weeks
  Interventions: Drug: PB-119 75ug
- PB-119 150ug (Experimental): PB-119 injection 150ug subcutaneously injected once-weekly for 12 weeks
  Interventions: Drug: PB-119 150ug
- PB-119 200ug (Experimental): PB-119 injection 200ug subcutaneously injected once-weekly for 12 weeks
  Interventions: Drug: PB-119 200ug
- placebo (Placebo Comparator): placebo injection subcutaneously injected once-weekly for 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PB-119 75ug — 60 eligible patients will be included in this group
  Arms: PB-119 75ug
Drug: PB-119 150ug — 60 eligible patients will be included in this group
  Arms: PB-119 150ug
Drug: PB-119 200ug — 60 eligible patients will be included in this group
  Arms: PB-119 200ug
Drug: placebo — 60 eligible patients will be included in this group
  Arms: placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel dose cohort, multiple dose study to evaluate the efficacy, safety, and tolerability of different doses of PB-119 in drug-naïve subjects with T2DM.

DETAILED DESCRIPTION:
Subjects will be assessed for eligibility over a 2-week screening period prior to a 2-week run-in period and a 12-week double-blind treatment period,4-week follow up period. The eligible patients will be randomized to 1 of 3 dose cohorts (A, B, or C). Each patient will subsequently be randomized within the designated cohort to active drug or placebo at a 3:1 active drug:placebo ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females between the ages of ≥18 and ≤70 years at Screening
2. Patients in whom T2DM has been diagnosed according to 1999 WHOT2DM diagnostic criteria
3. HbA1c ≥7.5% and ≤11% at Screening and at Week -1
4. Body mass index (BMI) ≥18.5 and ≤35.0 kg/m2 at Screening

Exclusion Criteria:

1. Female who is pregnant, intends to become pregnant or breast-feeding or is of child-bearing potential and not using adequate contraception methods throughout the trial
2. Treatment with any glucose lowing agent(s) within 3 months prior to screening.An exception is short-term treatment (no longer than 7 days in total) with insulin in connection with inter-current illness
3. Calcitonin ≥50 ng/L at screening
4. Patients with a personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia, type 2
5. Fasting triglyceride ≥500 mg/dL at Screening, or patients with a history of lipid disorders taking unstable treatment dosage (eg, statins) within 3 months prior to screening
6. Any acute or chronic condition that, in the opinion of the Investigator, would limit the patient's ability to complete and/or participate in this trial
7. Blood amylase or lipase >3x ULN, history of acute or chronic pancreatitis, or history of symptomatic gallbladder disease at Screening
8. Serum creatinine ≥1.5 mg/dL (male patients) or ≥1.4 mg/dL (female patients), or estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2 at Screening
9. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2x upper limit of normal (ULN) at Screening and pre-randomization
10. Severe cardiovascular diseases occurring within 6 months prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Change of glycosylated hemoglobin(HbA1c) | 12 weeks
  Change of HbA1c from baseline value to end of treatment

SECONDARY OUTCOMES:
Percentage of patients achieving HbA1c <7% | 12 weeks
  Percentage of patients achieving HbA1c <7% at Week 12
Percentage of patients achieving HbA1c ≤6.5% | 12 weeks
  Percentage of patients achieving HbA1c ≤6.5% at Week 12
HbA1c | 2, 4, and 8 weeks
  Changes of HbA1c from baseline value at Weeks 2, 4, and 8
Fasting plasma glucose(FPG) | 2, 4, 8, and 12 weeks
  Changes of fasting plasma glucose(FPG) from baseline value at Weeks 2, 4, 8, and 12.
2-hour postprandial glucose(2-h PPG) | 4, 8, and 12 weeks
  Changes of 2-hour postprandial glucose(2-h PPG) from baseline value at Weeks 4, 8, and 12.
Insulin | 4, 8, and 12 weeks
  Changes of insulin from baseline value at Weeks 4, 8, and 12
C-peptide | 4, 8, and 12 weeks
  Changes of C-peptide from baseline value at Weeks 4, 8, and 12
Self-monitoring of blood glucose (SMBG) | 4, 8, and 12 weeks
  Changes of mean profile and mean increments from baseline value of the 7-point SMBG

OTHER OUTCOMES:
Body mass index(BMI) | 2, 4, 8, and 12 weeks
  Changes of BMI from baseline value at Weeks 2, 4, 8, and 12.
Waist and hip circumferences and waist-to-hip ratio | 12 weeks
  Change of waist and hip circumferences and waist-to-hip ratio from baseline value at end of treatment(waist and hip circumferences will be used to calculate waist-to-hip ratio
Blood pressure(both systolic and diastolic) | 2, 4, 8, and 12 weeks
  Changes of blood pressure from baseline value at Weeks 2, 4, 8, and 12.
Blood lipid | 2, 4, 8, and 12 weeks
  Changes of blood lipid from baseline value at Weeks 2, 4, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, MD,PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

REFERENCES:
- [Derived] Ji L, Du Y, Xu M, Zhou X, Mo Z, Ma J, Li J, Li Y, Lin J, Wang Y, Yang J, Song W, Jin H, Pang S, Liu H, Li P, Liu J, Yao M, Li W, Jiang X, Shen F, Geng H, Zhou H, Ran J, Lei M, Du Y, Ye S, Guan Q, Lv W, Tan H, Chen T, Yang J, Qin G, Li S, Chen L. Efficacy and safety of PEGylated exenatide injection (PB-119) in treatment-naive type 2 diabetes mellitus patients: a Phase II randomised, double-blind, parallel, placebo-controlled study. Diabetologia. 2021 May;64(5):1066-1078. doi: 10.1007/s00125-021-05392-9. Epub 2021 Mar 9. PMID 33687487
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581